CLINICAL TRIAL: NCT01042262
Title: Maternal Oxygen Use During Delivery and Cord Blood Superoxide Dismutase: A Randomized Controlled Trial
Brief Title: Maternal Oxygen Use During Delivery and Cord Blood Superoxide Dismutase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Hany Aly, MD, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 120621
Record Dates: First submitted 2009-12-21; First posted 2010-01-05 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-12

CONDITIONS: Oxidative Stress; Fetal Distress
Keywords: Superoxide dismutase; Oxygen; Oxygen free radicals; Labor and delivery
MeSH Terms: conditions — Fetal Distress | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen Group (Experimental): Subjects received 100% oxygen via nasal cannula (flow =2 L/min)
  Interventions: Other: Oxygen
- Control Group (Placebo Comparator): Subjects were attached to a nasal cannula without any oxygen flow.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Oxygen — 100% Oxygen at a flow of 2 L/min
  Arms: Oxygen Group
Other: Placebo — No oxygen flow
  Arms: Control Group

SUMMARY:
When exposed to oxygen immediately after birth, newborns suffer from an oxidative stress with a significant decrease in serum concentration of the anti-oxidant enzyme superoxide dismutase. This oxidative stress has been consequently linked to the development of adverse outcomes in both premature and full term infants. In this study, we examined the effect of oxygen administration to delivering mothers immediately before and during labor on the newborn. In this randomized trial, we planned to measure superoxide dismutase in the umbilical cord blood when mothers received and did not receive oxygen..

DETAILED DESCRIPTION:
We conducted a prospective randomized controlled clinical trial on a cohort of delivering women who were admitted to the Childbirth center at the George Washington University Hospital. This study has been approved by the Institutional Review Board of the George Washington University and consents were obtained from all subjects before enrollment. All of the enrolled subjects met the following criteria: a) uncomplicated pregnancy, b) term gestational age from completed 37 weeks to 42 weeks, and c) normal spontaneous vaginal delivery (NSVD) or elective caesarean section. Pregnant women were excluded from this study if they had any of the following: a) hypertension, or eclampsia, b) pregnancy induced diabetes, c) anemia, d) other medical or surgical complications during the current pregnancy, e) rupture of amniotic membranes for more than 18 hours, f) history of infants with invasive group B Streptococcal disease in previous pregnancies, g) fetal distress before delivery and h) suspected chromosomal, and structural anomalies or congenital infections. We collected data on maternal history (age, race, parity and type of anesthesia) and birth history (anthropometric measurements, gestational age, sex, and Apgar scores).

Randomization: Once enrolled in the study, all of the subjects were randomly assigned to one of two groups using the sealed opaque envelopes technique. A nasal cannula was attached to all subjects and was connected to a flowmeter covered by a metal foil so that the managing obstetricians were not aware which group the particular subject belongs to. The Oxygen Group participants received 100% oxygen at 2 litters/minute starting at least 30 minutes before delivery. The Control Group participants had their nasal cannula still attached to a flowmeter that was turned off. Nasal cannula was disconnected from participants after delivery.

Monitoring procedure: Pregnant women were monitored continuously for heart rate, respiratory rate and oxygen saturation. If oxygen saturation decreased < 93% for at least 60 seconds, and/or when considered necessary by the obstetrician at any time, therapeutic oxygen was administered and the participant was excluded from the study.

Laboratory investigation: We obtained three samples of three mls of whole blood from each mother-infant pair in both groups. The first blood sample was obtained from the participants' peripheral vein at the time of enrollment before randomization (Baseline). The second blood sample was obtained from the placental side of umbilical cord after delivery. The third sample was obtained from the partcipants' peripheral vein within 4 hours after delivery.

We measured blood gases in each sample at the bedside using an iSTAT analyzer (Abbott, IL). The rest of the sample was used for SOD assays. It was collected in an iced-tube containing EDTA, and centrifuged at 4 ºC. Plasma was discarded and the erythrocyte suspension was washed with normal saline and centrifuged again twice. Washed erythrocyte suspensions were stored at -70 ºC until the time of assay.

SOD concentration was measured by an indirect colorimetric method using the highly water-soluble tetrazolium salt WST-1, which produces a water-soluble formazan dye upon reduction with a superoxide anion. The Cayman Chemical SOD assay kit was used for the measurement of SOD activity in erythrocyte lysate. SOD activity was assessed by measuring the dismutation of superoxide radicals generated by xanthine oxidize and hypoxanthine in a convenient 96 well format. This technique included a quality-controlled SOD standard. The standard curve, which was generated using this enzyme, provides a means to accurately quantify the activity of all three types of SOD (Cu/Zn-, Mn-, and Fe-SOD). SOD concentration expressed in IU per gram of hemoglobin content. Results of SOD concentration, pH, pCO2, pO2, base deficit, Ht and Na concentration were recorded.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated pregnancy
* term gestational age from completed 37 weeks to 42 weeks, and
* normal spontaneous vaginal delivery or elective caesarean section

Exclusion Criteria:

* hypertension, or eclampsia
* diabetes
* anemia
* other medical or surgical complications during the current pregnancy
* rupture of amniotic membranes for more than 18 hours
* history of infants with invasive group B Streptococcal disease in previous pregnancies
* fetal distress before delivery, and
* suspected chromosomal, and structural anomalies or congenital infections

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Superoxide dismutase concentration in umbilical cord blood | within 4 hours

SECONDARY OUTCOMES:
Superoxide dismutase concentration in maternal venous blood after delivery | within 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Nesterenko TH, Acun C, Mohamed MA, Mohamed AN, Karcher D, Larsen J Jr, Aly H. Is it a safe practice to administer oxygen during uncomplicated delivery: a randomized controlled trial? Early Hum Dev. 2012 Aug;88(8):677-81. doi: 10.1016/j.earlhumdev.2012.02.007. Epub 2012 Mar 23. PMID 22445187